CLINICAL TRIAL: NCT05517148
Title: Effects of an Immersive Virtual Reality Intervention Combined With Mindfulness-based Therapy on Mental Health in Nurses During the COVID-19 Pandemic: A Randomized Controlled Trial
Brief Title: Effects of an Immersive Virtual Reality Intervention Combined With Mindfulness-based Stress Reduction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Huichao Zhang, Professor, Nanjing University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: SJCX22_0701
Record Dates: First submitted 2022-08-23; First posted 2022-08-26 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Stress; COVID-19 Pandemic; Nurse's Role
Keywords: Mindfulness-based Stress Reduction; Virtual Reality; COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: The study utilized random sampling to recruit participants, and ethical approval was obtained prior to the commencement of the study. The participants were then divided into two groups through randomization, which was conducted by an independent researcher using the random number calculation procedure available at www.random.org. Following randomization, participants in the same department should were encouraged to adopt a unified intervention mode. Nurses working in the same department were assigned to the same group, and participants were not made aware of the existence of the other group existed. This form of masking is commonly used in randomised controlled trials to prevent potential bias from patients in the control group requesting the intervention or otherwise altering their behaviors. However, the investigators were aware of assignment. Before registering for this study, participants agreed to commence receiving the intervention in September 2022.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-based Stress Reduction by Therapeutic VR (Experimental): 47 participates were randomized and allocated to this treatment group. During the study, seven individuals were lost, and a total of 40 nurses participated in the final statistics. Of the seven individuals lost, two withdrew from the intervention due to personal reasons, while the remaining five terminated the intervention due to COVID-19 infection. The therapeutic intervention consisted of an eight-week group intervention that included the same amount of contact and meditations as MBT.
  Interventions: Device: Therapeutic VR
- Mindfulness-based Stress Reduction (Other): Received the same mindfulness therapy training audio as the other set, but did not watch the 3D scene on the VR device. At the end of the study, we will compensate them and let them use VR for relaxation training according to their wishes.
  Interventions: Device: Therapeutic VR

INTERVENTIONS:
Device: Therapeutic VR — Treatment module categories included: (1) Mindfulness-based stress reduction training: an audio conducting practice with breathing-based biofeedback training in immersive and interactive environments to support self-regulation and relaxation.
  Other Names: Mindfulness-based Stress Reduction

SUMMARY:
Mindfulness-based stress reduction (MBSR), a widely used method to improve mental state and sleep quality, was developed by Kabat-Zinn in 1970. The meditation of MBSR is effective in regulating patients' emotions, leading to reduced stress, pain, and psychological symptoms. Studies have demonstrated that MBSR has a positive impact on multiple psychological and physical symptoms in a variety of cancers. On this basis, investigators found that VR treatment can also help patients relax, and it has been widely used in cancer symptom relief in recent years. VR treatment involves using headset devices that fully restrict the vision field to content displayed inside the headset screen; As a treatment modality, VR provides a unique environment comprising 3D visually immersive experiences that are enriched with stereo sounds and elements such as rich colors and scenic environments that enhance elicitation of desired states of arousal and affect. Within the therapeutic context, VR may be flexibly designed and tailored to address the needs of specific conditions (eg, anxiety, depression, pain) auditory perception is not fully restricted, though the corresponding device-delivered auditory content commands attention.

DETAILED DESCRIPTION:
Recently, studies have revealed that individuals who have survived a COVID-19 infection may experience a range of persistent symptoms (Comelli et al., 2022; Nalbandian et al., 2021), indicating that the pandemic is far from over and its aftermath is difficult to eliminate completely. At the same time, the COVID-19 pandemic has presented unprecedented challenges for nurses around the world. Not only are they at the forefront of preventing and controlling the spread of the virus, but they are also the primary caregivers for patients experiencing the after-effects of the pandemic. Meanwhile, they also need to care for the patients with other illness. Some study evidence indicated that there is a shortage of nurses during the COVID-19 pandemic, and nursing staff are experiencing a high level of negative emotions (Jiang et al., 2022; Zhang et al., 2022).

The ongoing pandemic has had a huge impact on the mental health and work of nurses (Chen et al., 2021). Between 40% and 66.7% of surveyed health care workers reported mental health problems during the pandemic, according to a report by the OECD (Organisation for Economic Development and Cooperation, 2021). The stress caused by COVID-19 has contributed to workforce attrition, with many nurses opting to leave the profession (Organisation for Economic Development and Cooperation, 2021; World Health Organization, 2022). It has taken a heavy toll on the healthcare system. Maintaining the mental health of nurses is crucial. This is not only conducive to pandemic prevention and control, but also plays a significant role in the normal medical order.

ELIGIBILITY:
Registered nurses (RNs) working in target departments, working in target departments, including. The target departments mainly included internal medicine, surgical, emergency department, were included in this study. These nurses had direct contact with COVID-19 patients, making them more susceptible to experiencing negative mental health effects due to increased work pressure. Predefined exclusion criteria included serious carsickness reaction, psychological crisis with a definite diagnosis, and not being engaged in nursing work related to COVID-19. Nurse managers in different departments recommended participants for the study, and interested nurses were contacted to provide basic information and complete evaluation content. Recruitment took place in September 2022. We recorded the enrolled nurses, related basic information and outcome measures.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-09-25 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
The Hamilton Anxiety Rating Scale (HAM-A) | up to 8 weeks
  The HAM-A contains items, each scored on a 5-point scale (0, asymptomatic; 1, mild symptoms; 2, moderate symptoms; 3, severe symptoms; 4, extremely severe symptoms). The total sum score, ranging from 0 to 56, can be classified into four levels: 0, no anxiety symptoms; 1-17, mild anxiety; 18-24, moderate anxiety; 25-56, severe anxiety
Depression, anxiety, and stress scale (DASS-21) | up to 8 weeks
  The questionnaire of the Chinese version of DASS-21 comprises 21 items that assess three negative emotional experiences, namely depression, anxiety, and stress (Jiang et al., 2021). The depression factor consists of seven items (3, 5, 10, 13, 16, 17, 21), which are related to pathological dysthymia, low self-esteem, and low level of positive emotions. The anxiety factor comprises seven items (2, 4, 7, 9, 15, 19, 20), that related to the somatic and subjective experience of anxiety arousal. The stress factor includes seven items (1, 6, 8, 11, 12, 14, 18), that relate to negative emotionally. A 4-point score System was used (0=completely disagree, 1=partially agree, 2=mostly agree, 3=completely agree). Higher scores indicate stronger negative emotional experiences (Gomez et al., 2014; Oei et al., 2013).

SECONDARY OUTCOMES:
Work-related emotional score (WRE) | up to 8 weeks
  Nurses were asked to select a level of their mood at work during the COVID-19 to reflect their emotional attitude or degree of satisfaction towards work. The question posed was, "Has COVID-19 affected your mood at work?". The subjective scores range from 0 (no affected) to 10 (extremely affected).

CONTACTS AND LOCATIONS:
Overall Officials: Yuxi Zhang, master, Study Director — The First Affiliated Hospital with Nanjing Medical University
Locations (2):
- China (2):
  - siting YANG, Nanjing, Jiangsu
  - YANG Siting, Nanjing, Jiangsu

IPD SHARING:
Plan to Share IPD: No
Hope that the paper will be shared after it is accepted

REFERENCES:
- See also: Refer to related definitions — http://www.worldpediatricproject.org